CLINICAL TRIAL: NCT03960840
Title: Phase I/II, Open Label, Multicenter Study of Rapcabtagene Autoleucel in Adult Patients With CLL/SLL, 3L+ DLBCL, r/r ALL and 1L HR LBCL
Brief Title: Phase I/II Study of Rapcabtagene Autoleucel in CLL, 3L+ DLBCL, r/r ALL and 1L HR LBCL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYTB323A12101
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Diffuse Large B-cell Lymphoma; Acute Lymphoblastic Leukemia; Large B-cell Lymphoma
Keywords: CAR-T; Ibrutinib; CLL; DLBCL; ALL; BLRM; YTB323; Rapcabtagene autoleucel
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CLL/SLL (Experimental): Dose escalation of rapcabtagene autoleucel in combination with ibrutinib
  Interventions: Biological: Rapcabtagene autoleucel single agent; Drug: Ibrutinib
- 3L+ DLBCL (Experimental): Dose escalation and expansion of rapcabtagene autoleucel single agent in 3L+ DLBCL
  Interventions: Biological: Rapcabtagene autoleucel single agent
- Adult ALL (Experimental): Dose escalation of rapcabtagene autoleucel single agent in adult ALL
  Interventions: Biological: Rapcabtagene autoleucel single agent
- 1L HR LBCL (Experimental): Rapcabtagene autoleucel single agent in 1L HR LBCL
  Interventions: Biological: Rapcabtagene autoleucel single agent

INTERVENTIONS:
Biological: Rapcabtagene autoleucel single agent — Single infusion of rapcabtagene autoleucel
Drug: Ibrutinib — Tablets or capsules for oral daily use
  Arms: CLL/SLL

SUMMARY:
This is a phase I/II study to evaluate the feasibility, safety and preliminary antitumor efficacy of rapcabtagene autoleucel (also known as YTB323). Rapcabtagene autoleucel will be investigated in combination with ibrutinib in chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) and as single agent in diffuse large B-cell lymphoma (3L+ DLBCL), adult acute lymphoblastic leukemia (ALL) and 1st Line High Risk Large B-Cell Lymphoma (1L HR LBCL).

DETAILED DESCRIPTION:
This clinical trial is phase I/II open label, multi-center study of rapcabtagene autoleucel.

The Phase I part of the study comprises three independent treatment arms:

* Rapcabtagene autoleucel in combination with ibrutinib in adult CLL/SLL participants with SD or PR after at least 6 months of second or subsequent line ibrutinib therapy. As of 05-May-2021, this arm had completed enrollment.
* Rapcabtagene autoleucel single agent in adult DLBCL participants having failed two or more lines of chemotherapy and either having progressed (or relapsed) after autologous HSCT or being ineligible for or not consenting to the procedure.
* Rapcabtagene autoleucel single agent in adult relapsed/refractory ALL participants

The Phase II part of the study comprises two independent cohorts:

* Rapcabtagene autoleucel single agent in adult 3L + DLBCL participants having failed two or more lines of chemoimmunotherapy and either having progressed (or relapsed) after autologous HSCT or being ineligible for or not consenting to the procedure. This is an extension of the Phase I r/r DLBCL treatment arm to support Phase II objectives
* Rapcabtagene autoleucel single agent in newly diagnosed, adult 1L HR LBCL participants defined as IPI 3-5 and/or DH/TH disease who have completed 2 cycles of CIT and have a response of PR/SD (with a Deauville score of 4-5).

In the Phase I part of the trial, the 3L+ DLBCL and ALL arms consist of two parts: a dose escalation part to evaluate feasibility, characterize safety and identify the recommended dose (RD) of rapcabtagene autoleucel, and may be followed by a dose expansion part to further characterize safety, study rapcabtagene autoleucel cellular kinetics and assess preliminary antitumor activity. Once the RD of rapcabtagene autoleucel is determined for each arm, the corresponding expansion part may commence.

In the Phase II part of the trial, approximately 70 additional participants will be enrolled in a 3L+ DLBCL cohort treated at the recommended dose (RD). Including the 3L+ DLBCL participants who were treated at the RD from the Phase I part, it is planned to have in total a cohort of approximately 100 participants included in the primary efficacy analysis based on the efficacy analysis set. In addition, a separate cohort in 1LHR LBCL will be included, with approximately 50-60 participants planned for the primary efficacy analysis based on the efficacy analysis set.

Participants will be followed under the current treatment protocol for safety and efficacy within this trial for a minimum of 2 years before being transferred to the long-term follow-up trial. Once the study is complete, participants will be enrolled in a post-study long term follow-up for lentiviral vector safety for up to 15 years. This post-study long term follow-up for lentiviral vector safety will continue under a separate destination protocol.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-1 for ALL and DLBCL
* ECOG performance status 0-2 for 1L HR LBCL at screening
* CLL or SLL diagnosis according to iwCLL criteria
* CLL/SLL in SD or PR after at least 6 months of ibrutinib, either as second or subsequent line of therapy
* DLBCL diagnosis by local histopathology
* DLBCL relapsed or refractory after 2 or more lines of therapy, including autologous hematopoietic stem cell transplantation (HSCT)
* Refractory or relapsed CD19-positive ALL
* ALL with morphologic disease in the bone marrow

  1L HR LBCL - Considered to be high-risk based on at least 1 of the following at diagnosis:
  * IPI score of 3, 4 or 5
  * MYC and BCL2 and/or BCL6 rearrangement (DH/TH lymphoma)
* Participants must have received 2 cycles of frontline therapy for LBCL with R-CHOP or Pola-R-CHP or DA-EPOCH-R. Participants with DH/TH lymphoma must have received at least one cycle (the most recent) DA-EPOCH-R.
* Participants must have a positive PET per Lugano classification (Deauville PET score of 4 or 5 and an overall response of PR/SD) after 2 cycles of frontline CIT. Note: Patient's with Deauville PET score of 5 and overall response of PD, or with Deauville PET score of 1, 2, or 3 and overall response of CR, are not eligible for this trial.

Exclusion Criteria:

* Prior CD19-directed therapy
* Prior administration of a genetically engineered cellular product
* Prior allogeneic HSCT
* Richter's transformation

  * For 1L HR LBCL: Richter's transformation, Burkitt lymphoma, primary DLBCL of CNS, DLBCL associated with chronic inflammation, intravascular large B-cell lymphoma, ALK- positive large B-cell lymphoma, HHV8 positive LBCL, DLBCL leg type or EBV positive DLBCL, NOS.
* Active CNS lymphoma

  * For 1L HR LBCL: Active or prior history CNS involvement by malignancy
* Targeted small molecule or kinase inhibitor within 2 weeks from leukapheresis

Other protocol-defined inclusion/exclusion may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose recommendation: Incidence and nature of Dose Limiting Toxicities (Dose Escalation part only) | 28 days
Phase 1: Safety: Incidence and severity of AEs and SAEs, including changes in laboratory values, ECG and vital signs | 24 months
Phase 1: Tolerability: Ibrutinib dose modifications in the CLL/SLL arm | 24 months
Phase 1: Manufacture success: Number of patients infused with planned target dose | 24 months
Phase 2: Complete Response Rate (CRR) as assessed by local Investigator | 24 months
  CRR defined as best overall response (BOR) of CR after rapcabtagene autoleucel infusion as per Lugano criteria for 3L+ Diffuse Large B-Cell Lymphoma (DLBCL) and 1L High Risk Large B-Cell (HR LBCL)

SECONDARY OUTCOMES:
Phase 1: Complete Response (CR)/Partial Response (CR) in CLL/SLL | 24 months
  per international workshop on Chronic Lymphocytic Leukemia (iwCLL) response criteria
Phase 1: BOR of CR/PR per Lugano criteria in 3L+ DLBCL | 24 months
Phase 1: Duration of response (DOR) in CLL/SLL and 3L+ DLBCL | 24 months
  DOR as assessed by time from first achievement of CR/PR after rapcabtagene autoleucel infusion until first documented disease progression or death due to any cause
Phase 1: BOR in ALL as assessed by an Independent Review Committee (IRC) | month 3
  BOR of CR/CRi by 3 months after rapcabtagene autoleucel infusion as per IRC assessment.
Phase 1: DOR in ALL as assessed by an Independent Review Committee | 24 months
  DOR, defined as the time from achievement of CR or CRi to relapse or death due to any cause
Phase 1: EFS in ALL as assessed by an Independent Review Committee | 24 months
  EFS, defined as the date from rapcabtagene autoleucel infusion to the earliest date of relapse after CR/CRi, treatment failure (defined as failure to achieve CR/CRi within 12 weeks of infusion), or death due to any cause
Phase 1: BOR in ALL as assessed by local Investigator | 24 months
  BOR of CR/CRi
Phase 1: DOR in ALL as assessed by local Investigator | 24 months
  DOR, defined as the time from achievement of CR or CRi to relapse or death due to any cause.
Phase 1: EFS in ALL as assessed by local Investigator | 24 months
  EFS, defined as the date from rapcabtagene autoleucel infusion to the earliest date of relapse after CR/CRi, treatment failure (defined as failure to achieve CR/CRi within 12 weeks of infusion), or death due to any cause
Phase 1: Overall survival in adult ALL | 24 months
  OS defined as time from the date of infusion to the date of death due to any reason
Phase 1: MRD negative status by flow cytometry in adult ALL | 24 months
Phase 1: Quality of life in adult ALL patients enrolled in the expansion part by use of Electronic Patient Reported Outcomes (ePRO) as per EORTC QLQ-C30 questionnaire | 24 months
Phase 1: Quality of life in adult ALL patients enrolled in the expansion part by use of Electronic Patient Reported Outcomes (ePRO) as per EQ-5D-3 questionnaire | 24 months
Phase 1/2: Cellular kinetics | 24 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in peripheral blood, bone marrow and lymph nodes
Phase 1/2: Immunogenicity | 24 months
  Cellular and humoral responses to the CAR transgene
Phase 2: Overall response rate (ORR) | 24 months
  ORR defined as BOR of CR/PR as per Lugano criteria in 3L+ DLBCL and 1L HR LBCL
Phase 2: Complete Response Rate (CRR) | months 3, 6
  CRR at months 3, 6 in 3L+ DLBCL
Phase 2: Complete Response Rate (CRR) | months 6, 12
  CRR at months 6, 12 in 1L HR LBCL
Phase 2: Duration of response (DOR) | 24 months
  DOR defined as time from first CR/PR to first documented progression or death due to any cause in 3L+ DLBCL and 1L HR LBCL
Phase 2: Progression-free survival (PFS) | 24 months
  PFS defined as time from rapcabtagene autoleucel infusion to first documented progression or death due to any cause in 3L+ DLBCL and 1L HR LBCL
Phase 2: Event-free survival (EFS) | 24 months
  EFS defined as time from rapcabtagene autoleucel infusion to first documented progression, start of new anti-lymphoma therapy, biopsy-proven residual disease on or after month 6, or death due to any cause in 1L HR LBCL
Phase 2: Overall survival (OS) | 24 months
  OS defined as time from date of rapcabtagene autoleucel infusion to date of death due to any cause in 3L+ DLBCL and 1L HR LBCL
Phase 2: Complete Response Rate (CRR) in subgroups 1) IPI 4-5 or DH/TH and 2) IPI 3 and not DH/TH | months 6, 12
  CRR at months 6, 12 in 1L HR LBCL
Phase 2: Overall response rate (ORR) in subgroups 1) IPI 4-5 or DH/TH and 2) IPI 3 and not DH/TH | 24 months
  ORR defined as BOR of CR/PR as per Lugano criteria 1L HR LBCL
Phase 2: Duration of response (DOR) in subgroups 1) IPI 4-5 or DH/TH and 2) IPI 3 and not DH/TH | 24 months
  DOR defined as time from first CR/PR to first documented progression or death due to any cause in 1L HR LBCL
Phase 2: Progression-free survival (PFS) in subgroups 1) IPI 4-5 or DH/TH and 2) IPI 3 and not DH/TH | 24 months
  PFS defined as time from rapcabtagene autoleucel infusion to first documented progression or death due to any cause in 1L HR LBCL
Phase 2: Event-free survival (EFS) in subgroups 1) IPI 4-5 or DH/TH and 2) IPI 3 and not DH/TH | 24 months
  EFS defined as time from rapcabtagene autoleucel infusion to first documented progression, start of new anti-lymphoma therapy, biopsy-proven residual disease on or after month 6, or death due to any cause in 1L HR LBCL
Phase 2: Overall survival (OS) in subgroups 1) IPI 4-5 or DH/TH and 2) IPI 3 and not DH/TH | 24 months
  OS defined as time from date of rapcabtagene autoleucel infusion to date of death due to any cause in 1L HR LBCL
Phase 2: Manufacturing vein to door time | 24 months
  Time from apheresis completion until return of rapcabtagene autoleucel product to the clinic or hospital

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (11):
  - University of California LA, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Uni of Chi Medi Ctr Hema and Onco, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Mass Gen Hosp Cancer Center, Boston, Massachusetts
  - University of Pennsylvania Clinical, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - St Davids South Austin Medical Ctr, Austin, Texas
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Vienna, Austria
- France (4):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rennes
- Germany (3):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Essen
- Italy (4):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Japan (3):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Fukuoka
- Spain (8):
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia

IPD SHARING:
Plan to Share IPD: No